CLINICAL TRIAL: NCT03922542
Title: Randomized Comparison of Standard vs. Accelerated Corneal Crosslinking for Treatment of Progressive Keratoconus or Ectasia
Brief Title: Comparison of Standard vs. Accelerated Corneal Crosslinking
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-003
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Keratoconus; Ectasia Corneal
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated (Active Comparator): Treatment with 0.1% riboflavin eye drops and 9 mW/cm2 UVA light for 10 minutes
  Interventions: Combination Product: riboflavin 0.1%
- Standard (Active Comparator): Treatment with 0.1% riboflavin eye drops and 3 mW/cm2 UVA light for 30 minutes
  Interventions: Combination Product: Riboflavin 0.1%

INTERVENTIONS:
Combination Product: riboflavin 0.1% — Use of riboflavin 0.1% eye drops and 9 mW/cm2 UVA light for 10 minutes
  Arms: Accelerated
Combination Product: Riboflavin 0.1% — Use of riboflavin 0.1% eye drops and 3 mW/cm2 UVA light for 30 minutes
  Arms: Standard

SUMMARY:
The study objective is to compare accelerated and standard corneal crosslinking for treatment of progressive keratoconus or corneal ectasia.

ELIGIBILITY:
Inclusion Criteria:

* Documented keratoconus or ectasia after refractive surgery

Exclusion Criteria:

* Insufficient corneal thickness
* Ocular condition that may predispose the eye to complications
* History of chemical injury or delayed epithelial healing
* Condition that would interfere with or prolong epithelial healing
* Known sensitivity to treatment medications
* Pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximum keratometry | 6 months
  assessed by corneal tomography

SECONDARY OUTCOMES:
Change in corrected distance visual acuity | 6 months
  assessed with Snellen chart
Change in uncorrected distance visual acuity | 6 months
  assessed with Snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price MO, Fairchild K, Feng MT, Price FW Jr. Prospective Randomized Trial of Corneal Cross-linking Riboflavin Dosing Frequencies for Treatment of Keratoconus and Corneal Ectasia. Ophthalmology. 2018 Apr;125(4):505-511. doi: 10.1016/j.ophtha.2017.10.034. Epub 2017 Dec 2. PMID 29203068
- [Background] Lautert J, Doshi D, Price FW Jr, Price MO. Corneal Epithelial Remodeling After Standard Epithelium-off Corneal Cross-linking in Keratoconic Eyes. J Refract Surg. 2018 Jun 1;34(6):408-412. doi: 10.3928/1081597X-20180402-03. PMID 29889294
- [Background] Price MO, Feng MT, Price FW Jr. Patient satisfaction with epithelium-off corneal crosslinking. J Cataract Refract Surg. 2018 Mar;44(3):323-328. doi: 10.1016/j.jcrs.2017.12.023. Epub 2018 Mar 28. PMID 29605283